CLINICAL TRIAL: NCT05206708
Title: Assesment of the Efficacy of Personalized Parent-child Psychotherapy Evaluating Symptoms in Children Under 3 Years Old and Parent-child Interaction.
Brief Title: Assesment of the Efficacy of Personalized Parent-child Psychotherapy in Children Under 3 Years Old
Acronym: ECRIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/484
Record Dates: First submitted 2022-01-10; First posted 2022-01-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Child Behavior Disorders; Parent-Child Relations
MeSH Terms: conditions — Child Behavior Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: 117 dyads will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (Active Comparator): Standard psychodynamic therapy
  Interventions: Behavioral: Standard of care
- Personalized care (Experimental): Psychodynamic therapy or interactive guidance therapy
  Interventions: Behavioral: Personalized psychotherapy

INTERVENTIONS:
Behavioral: Personalized psychotherapy — Strategy including personalized psychotherapy
  Arms: Personalized care
Behavioral: Standard of care — Strategy based standard intregrative psychodynamic therapy
  Other Names: Standard intregrative psychodynamic therapy
  Arms: Standard care group

SUMMARY:
This study aims to assess the efficacy at 4 months of a personalized strategy comparatively to a standard Psychodynamic Integrative Therapy, on childrens' symptom improvment

DETAILED DESCRIPTION:
3 evaluations are performed: before treatment, at the end of the treatment and one year after the treatment.

evaluations include assessment of: children's symptom parent-infant interaction quality parental competencies parental perception of the child by his/her parent parent-therapist alliance hair cortisol concentration

ELIGIBILITY:
Inclusion Criteria:

* Families who are requesting a consultation for functional or behavioural problems of their child
* Children under the age of 3

Exclusion Criteria:

* Parents suffering from a severe untreated psychiatric disorder
* Difficulties in speaking French
* Children with Autistic spectrum disorder
* Families already in care

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of therapy | Month 4
  To assess the efficacy at 4 months of a personalized strategy by Interactive Guidance or Psychodynamic Therapy, comparatively to a standard Psychodynamic Therapy, on child symptoms assessed with the "Symptom Check List"

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane Coady-Vulliez, MD, Principal Investigator — CHU Besançon
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - CHU de Montpellier, Montpellier
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - CHU de Reims, Reims

IPD SHARING:
Plan to Share IPD: No